CLINICAL TRIAL: NCT01463137
Title: Computerized Attention Bias Modification Training in Social Phobia/Social Anxiety Disorder
Brief Title: Attention Bias Modification Training in Social Phobia/Social Anxiety Disorder
Acronym: SOFIE-11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Per Carlbring, PhD, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOFIE-11
Record Dates: First submitted 2011-10-27; First posted 2011-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Social Phobia
Keywords: social phobia; anxiety
MeSH Terms: conditions — Phobia, Social; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Control training with words (Sham Comparator): Computerized, internet-based control training program. Participant is exposed to a pair of words -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words and is then asked to press the corresponding arrow button on a keyboard. A total of 192 word pairs are shown during a session. One third is neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe follows the more positive word and the more negative word with equal frequency.
  Interventions: Behavioral: Attention bias modification
- Control training with words + pictures (Sham Comparator): Computerized, internet-based control training program. Participant is exposed to a pair of words or a pair of faces -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words or faces and is then asked to press the corresponding arrow button on a keyboard. A total of 96 word pairs and 96 face pairs are shown during a session. One third is neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe follows the more positive stimulus and the more negative stimulus with equal frequency.
  Interventions: Behavioral: Attention bias modification
- Positive bias training with words (Active Comparator): Computerized, internet-based training program for implicit modification of cognitive bias of attention, variant 1. Participant is exposed to two words -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words and is then asked to press the corresponding arrow button on a keyboard. A total of 192 word pairs are shown during a session, of one third is the neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe always follows the more positive word.
  Interventions: Behavioral: Attention bias modification
- Positive bias training with words + pictures (Active Comparator): Computerized, internet-based training program for implicit modification of cognitive bias of attention, variant 2. Participant is exposed to a pair of words or a pair of faces -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words or faces and is then asked to press the corresponding arrow button on a keyboard. A total of 96 word pairs and 96 face pairs are shown during a session. One third is neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe always follows the more positive word or face.
  Interventions: Behavioral: Attention bias modification
- Negative bias training with words (Active Comparator): Computerized, internet-based training program for implicit modification of cognitive bias of attention, variant 3. Participant is exposed to two words -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words and is then asked to press the corresponding arrow button on a keyboard. A total of 192 word pairs are shown during a session. One third is neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe always follows the more negative word.
  Interventions: Behavioral: Attention bias modification
- Negative bias training with words + pictures (Active Comparator): Computerized, internet-based training program for implicit modification of cognitive bias of attention, variant 4. Participant is exposed to a pair of words or a pair of faces -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words or faces and is then asked to press the corresponding arrow button on a keyboard. A total of 96 word pairs and 96 face pairs are shown during a session. One third is neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe always follows the more negative word or face.
  Interventions: Behavioral: Attention bias modification

INTERVENTIONS:
Behavioral: Attention bias modification — All arms will consist of 10 minutes of training in front of a computer screen (192 trials) once a day for 14 days.

SUMMARY:
A study investigating six different versions of a computerized attention bias modification internet program in the treatment of social phobia / social anxiety disorder.

DETAILED DESCRIPTION:
Previous studies have shown that individuals with social phobia have attention biases, often focusing on aversive stimuli or avoiding aversive stimuli. Computerized training programs have been developed to implicitly direct the users attention towards a neutral, non-threatening stimuli. In this study, such a program will be compared with a program that implicitly directs the users' attention towards threatening cues. Pre/post-measurements will be compared in a sample of individuals that meet diagnostic criteria of Social Anxiety Disorder. Participants will be randomized to one of three groups, receiving one of the two variants of the attention bias modification program or a control training program.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet criteria for social phobia using the International classification system Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV).
* Comorbidity is allowed, but social phobia must be the primary diagnosis.

Exclusion Criteria:

* Below 18 years old.
* Individuals who are suicide prone will be excluded from the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Liebowitz Social Anxiety Scale self rated version | pretreatment (week 0), post treatment (week 2), 4 month follow-up
  Change from baseline in social anxiety symptoms expected between time frames.

SECONDARY OUTCOMES:
Change from baseline in Social Phobia Screening Questionnaire | Pretreatment (week 0), post treatment (week 2), 4 month follow-up
  Social Phobia Screening Questionnaire (SPSQ), diagnostic tool for social phobia.
  Change from baseline in social anxiety symptoms expected between time frames.
Change from baseline in Social Interaction Anxiety Scale (SIAS) | Pretreatment (week 0), post treatment (week 2), 4 month follow-up
  Change from baseline in social anxiety symptoms expected between time frames.
Change from baseline in Social Phobia Scale (SPS) | Pretreatment (week 0), post treatment (week 2), 4 month follow-up
  Change from baseline in social anxiety symptoms expected between time frames.
Change from baseline in Montgomery Åsberg Depression Rating Scale (MADRS-S) | Pretreatment (week 0), post treatment (week 2), 4 month follow-up
  Measure depression.
  Change from baseline in depressive symptoms expected between time frames.
Change from baseline in Quality of Life Inventory (QOLI) | Pretreatment (week 0), post treatment (week 2), 4 month follow-up
  Measure quality of life.
  Change from baseline in quality of life expected between time frames.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Umeå University, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Result] Boettcher J, Leek L, Matson L, Holmes EA, Browning M, MacLeod C, Andersson G, Carlbring P. Internet-based attention bias modification for social anxiety: a randomised controlled comparison of training towards negative and training towards positive cues. PLoS One. 2013 Sep 30;8(9):e71760. doi: 10.1371/journal.pone.0071760. eCollection 2013. PMID 24098630